CLINICAL TRIAL: NCT05202717
Title: Construction of the Early Warning and Prevention System for Urinary Incontinence in the Elderly--the Effect of a New Type of Pelvic Floor Rehabilitation Device PHENIX U4+ on the Treatment of Urinary Incontinence--a Multi-center Randomized Controlled Clinical Study
Brief Title: the Effect of a New Type of Pelvic Floor Rehabilitation Device PHENIX U4+ on the Treatment of Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Xiuli, Chief Gynecology Physician, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PkuH5
Record Dates: First submitted 2021-11-23; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-10

CONDITIONS: Urinary Incontinence
Keywords: new type of pelvic floor rehabilitation device PHENIX U4+; Traditional pelvic floor electrical stimulation therapy instrument
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PHENIX U4+ (Experimental): Electrical stimulation treatment for patients with urinary incontinence using a new type of pelvic floor therapy instrument
  Interventions: Device: PHENIX U4+
- Traditional pelvic floor electrical stimulation therapy instrument (Active Comparator): Electrical stimulation treatment for patients with urinary incontinence using traditional pelvic floor therapy instrument
  Interventions: Device: Traditional pelvic floor treatment instrument

INTERVENTIONS:
Device: PHENIX U4+ — The newly developed domestic PHENIX U4+ is relatively small in size. In addition to the smooth muscle stimulation function of the traditional therapy device, its electrical stimulation waveform setting can also stimulate the striated muscle, and adds more than 10 A3 reflex treatment options, which can inhibit Urinary reflex, resulting in symptoms related to urinary incontinence in the patient.
  Arms: PHENIX U4+
Device: Traditional pelvic floor treatment instrument — Traditional pelvic floor treatment instrument commonly used in clinical practice
  Arms: Traditional pelvic floor electrical stimulation therapy instrument

SUMMARY:
Enrolled patients with urinary incontinence in Peking University People's Hospital, Wuhan People's Hospital, Zhongshan People's Hospital, and Jiangsu Maternity and Child Health Hospital in the Department of Gynecology, and collected baseline data. The random number table was used to divide the period into observation group and control group. The observation group was treated with a new type of pelvic floor rehabilitation therapy device PHENIX U4+, and the control group was treated with a traditional pelvic floor electrical stimulation therapy device. Follow-up observations during the treatment period and at the end of the treatment, 3 months and 6 months, the main follow-up content includes 1h pad test, 72-hour urination diary, modified Oxford muscle strength classification diagnosis, urinary incontinence-related questionnaires, new equipment inspections, etc. , Track and compare the treatment effect.

DETAILED DESCRIPTION:
Use two pelvic floor treatment devices to treat urinary incontinence, collect relevant questionnaires and pelvic floor muscle strength, and compare the two treatment devices.

ELIGIBILITY:
Inclusion Criteria:1) 18 years old and above; 2) Have a history of sexual life; 3) Plan to live locally for a long time; 4) Mild to moderate pressure, urgency or mixed urinary incontinence; 5) The patient agrees to conduct the study and signs an informed consent form.

Exclusion Criteria:

1. Combined pelvic organ prolapse (with extrahymen bulging);
2. Obesity (BMI>28kg/m2, BMI=weight (kg)/height square (m2));
3. Uncontrolled asthma and chronic obstructive pulmonary disease (COPD);
4. Combined connective tissue disease;
5. Women with unclean lochia during pregnancy, within 6 weeks of postpartum and postpartum
6. Malignant tumors;
7. Combined neurological diseases (patients with epilepsy and dementia);
8. Those with a synchronized pacemaker on their chest (biofeedback can be done).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The difference in the effective rate of urinary incontinence treatment between the two groups | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
  The effective rate of urinary incontinence treatment is judged by whether it leaks urine or not

SECONDARY OUTCOMES:
Differences in pelvic floor electromyography between the two groups | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
Differences in 72-hour urination diary | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
  reflect urination of 72 hours
Person coefficient of correlation between results of gynecological examination and new equipment examination | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
Differences in questionnaire score： PFDI-20 | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
  Questionnaires reflecting pelvic floor function, lower urinary tract symptoms, and quality of life
Differences in questionnaire score： ICI-Q-SF | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
  Questionnaires reflecting lower urinary tract symptoms
Differences in questionnaire score： OABSS | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
  Questionnaires reflecting lower urinary tract symptoms
Differences in questionnaire score： UDI-6 | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
  Questionnaires reflecting lower urinary tract symptoms, and quality of life
Differences in pelvic floor pressure test between the two groups | Before treatment, immediately after treatment, three months after treatment, and six months after treatment
Differences in pelvic floor tension test between the two groups | Before treatment, immediately after treatment, three months after treatment, and six months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 1 year